CLINICAL TRIAL: NCT07222553
Title: Open-label, Uncontrolled, Multicenter Trial to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Inebilizumab in Children From 2 Years to Less Than 18 Years of Age With Immunoglobulin G4-related Disease (IgG4-RD)
Brief Title: Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Inebilizumab in Pediatric Participants With IgG4-RD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240202; 2025-520988-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Immunoglobulin G4-related Disease
Keywords: Immunoglobulin G4-related Disease; Inebilizumab; AMG 335; IgG4-related disease; IgG4-RD
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inebilizumab (Experimental): Participants will receive Inebilizumab via intravenous (IV) infusion.
  Interventions: Drug: Inebilizumab

INTERVENTIONS:
Drug: Inebilizumab — Inebilizumab will be administered via IV infusion.

SUMMARY:
The primary objectives of this study are to characterize the pharmacokinetics (PK) and pharmacodynamics (PD), as well as to assess the safety and tolerability, of inebilizumab in pediatric participants with IgG4-RD.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must weigh ≥ 17 kg to be eligible for enrollment.
2. Participant has provided informed consent/assent before initiation of any study-specific activities/procedures. Participant's legally authorized representative has provided informed consent when the participant is legally too young to provide informed consent, and the participant has provided written assent based on local regulations and/or guidelines before any study-specific activities/procedures being initiated.
3. Age 2 to < 18 years at the time of screening. For participants who reach the age of legal consent during the clinical study, notification will be required, and a new consent form must be signed by the participant for continuation in the study.
4. Clinical diagnosis of IgG4-RD.
5. Fulfillment of the 2019 American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) classification criteria as determined by the principal investigator (PI) at screening. Specifically, participants must meet the classification criteria entry requirements (including involvement of one of the following organs: pancreas, bile ducts/biliary tree, orbits, lungs, kidneys, lacrimal glands, major salivary glands, retroperitoneum, aorta, pachymeninges, or thyroid gland [Riedel's thyroiditis]), must not meet any of the classification criteria exclusions, and must achieve at least 20 classification criteria inclusion points.
6. Receipt of all age-appropriate and locally-required vaccinations before screening.
7. Participants requiring treatment in addition to or other than glucocorticoids (GCs) for IgG4-RD according to PI's assessment at screening.
8. Participants who are on GCs for the treatment of IgG4-RD should remain on a stable dose for at least 2 weeks before enrollment (Day 1). Tapering post enrollment will be at PI's discretion.

Key Exclusion Criteria:

1. Participants with any of the following abnormal liver function tests in the presence of hepatobiliary IgG4-RD activity:

   * aspartate aminotransferase (AST) > 10 × upper limit of normal (ULN)
   * alanine aminotransferase (ALT) > 10 × ULN
   * total bilirubin (TBL) > 5 × ULN Screening liver function tests may be repeated before Day 1 to permit abnormal values due to hepatobiliary IgG4-RD activity to respond to GC treatment.
2. Evidence of significant hepatic, renal, or metabolic dysfunction or significant hematological abnormality, including any of the following at screening (one repeat test may be conducted to confirm results within the same screening period):

   * platelet count < 75000/μL (or < 75 × 109/L)
   * absolute neutrophil count < 1200 cells/μL
   * total Ig < 600 mg/dL
   * CD4 T lymphocyte count < 300 cells/µL
   * hemoglobin < 8 g/dL (or < 80 g/L).
3. Estimated glomerular filtration rate < 45 mL/min/1.73 m^2.
4. B-cell counts < one-half of the lower limit of normal (LLN) for age according to the central laboratory.
5. Diagnosed with a concurrent autoimmune disease that is uncontrolled or requires any prohibited medication (unless approved by the medical monitor).
6. Clinically significant serious active or chronic viral, bacterial, or fungal infection that requires treatment with anti-infectives, hospitalization, or, in the investigator's opinion, represents an additional risk to the participant, within 2 months before Day 1 of study.
7. Known history of congenital or acquired immunodeficiency (eg, due to human immunodeficiency virus [HIV] infection, splenectomy, immunosuppression-related or idiopathic T-cell deficiencies) that predisposes the participant to infection.
8. Positive test for chronic hepatitis B infection at screening, defined as either: (1) Positive hepatitis B surface antigen (HBsAg); or (2) Positive hepatitis B core antibody (anti-HBc) PLUS negative hepatitis B surface antibody (anti-HBs). Note: Participants with a positive anti-HBs only, or a positive anti-HBc plus positive anti-HBs and negative HBsAg, are eligible to enroll.
9. Receipt of any of the following before Day 1: alemtuzumab, total lymphoid irradiation, bone marrow transplant, T-cell vaccination therapy.
10. Receipt of any of the following within 2 months before Day 1: azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, cyclophosphamide, tocilizumab, satralizumab, eculizumab, and mitoxantrone.
11. Receipt of rituximab or any experimental B-cell depleting agent (eg, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab), or any non-depleting B-cell-directed therapy (eg, belimumab), abatacept, within 6 months before screening unless B-cell counts have returned to ≥ one-half the LLN.
12. Receipt of any live or attenuated vaccine (administration of inactivated [killed] vaccine is acceptable) within 4 weeks before Day 1, Bacillus Calmette-Guérin vaccine within 1 year of screening, or blood transfusion within 4 weeks before screening or during screening.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-04-03 (Estimated); Primary Completion 2031-06-10 (Estimated); Study Completion 2031-06-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Inebilizumab | Up to Day 561
Area Under the Plasma Concentration-time Curve (AUC) of Inebilizumab | Up to Day 561
Clearance (CL) of Inebilizumab | Up to Day 561
Terminal Half-life (t½) of Inebilizumab | Up to Day 561
Volume of Distribution at Steady-state (Vss) of Inebilizumab | Up to Day 561
Change from Baseline in CD20+ B-cell Counts | Baseline and Day 561
Number of Participants Experiencing Adverse Events (AEs) | Up to Day 561
Number of Participants Experiencing Serious Adverse Events (SAEs) | Baseline up to Day 561
Number of Participants Experiencing Events of Interest (EOIs) | Baseline up to Day 561
Number of Participants Experiencing Clinically Significant Changes from Baseline in Laboratory Parameters | Baseline up to Day 561
Number of Participants Experiencing Clinically Significant Changes from Baseline in Vital Signs | Baseline up to Day 561

SECONDARY OUTCOMES:
Time-to-first Treated Flare Across 52 Weeks | Up to Week 52
Percentage of Flare-free Participants Across 52 Weeks | Up to Week 52
Annualized Flare Rate Across 52 Weeks | Up to Week 52
Presence of Antidrug Antibodies (ADA) Before and After Initiation of Treatment | Day 1 to Day 561
Percent Reduction from Baseline in Daily Glucocorticoid Dose at Week 52 | Baseline and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com